CLINICAL TRIAL: NCT01738308
Title: Investigating the Effect of Healing Touch on Post-Operative Recovery of Pediatric Tonsillectomies and Adenoidectomies Patients Ages 3 & 4
Brief Title: The Effects of Healing Touch on Post Operative Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: American Holistic Nurses Association (AHNA) (Unknown); Carolyn Stoll Research Fund (Cincinnati Childrens Hospital) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2011-1572
Record Dates: First submitted 2012-11-28; First posted 2012-11-30 (Estimated); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Surgery; Stress; Pain; Children; Post-Traumatic Stress Disorder
Keywords: Healing Touch; Pediatrics; surgery; stress; pain; Pediatric Stress; maladaptive behaviors; energy medicine; emergence delirium; emergence agitation; length of stay; ease of wake up; distress parents; distress pediatric patients; Pediatric Post-Traumatic Stress Disorder
MeSH Terms: conditions — Pain; Stress Disorders, Post-Traumatic; Emergence Delirium | interventions — Touch; Therapeutic Touch; Presenteeism

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healing Touch Treatment (Experimental): Healing Touch Treatment
  When enter PACU + usual standard of care.
  The Healing Touch practitioner will be at the bedside when the patient is first brought to the PACU. The HT practitioner will center and then attune with the child, connecting their energy with the child and setting the intention for healing for the child's highest good. The practitioner will then place one hand on the center of the patient's chest in the "high heart" area. The practitioner will hold this position until they feel a deep connection and "quieting" within the patient's energy. When the patient is awake and parents have been called to the bedside the HT practitioner will energetically ground and release the patient,
  Interventions: Procedure: Healing Touch
- Sham Healing Touch Treatment (Sham Comparator): Usual standard of post operative care plus a sham Heal Touch treatment upon entering the post anesthesia care unit. Treatment done by untrained study staff using same hand locations.
  Interventions: Procedure: Healing Touch Sham Treatment
- Control- No treatment done (No Intervention): Usual standard of post operative care with no additional intervention

INTERVENTIONS:
Procedure: Healing Touch — When enter PACU + usual standard of care.
  The Healing Touch practitioner will be at the bedside when the patient is first brought to the PACU. The HT practitioner will center and then attune with the child, connecting their energy with the child and setting the intention for healing for the child's highest good. The practitioner will then place one hand on the center of the patient's chest in the "high heart" area. The practitioner will hold this position until they feel a deep connection and "quieting" within the patient's energy. When the patient is awake and parents have been called to the bedside the HT practitioner will energetically ground and release the patient,
  Other Names: Energy Therapy; Reiki
  Arms: Healing Touch Treatment
Procedure: Healing Touch Sham Treatment — The untrained in energy work study staff will be at the bedside when the patient is first brought to the PACU. The practitioner will then place one hand on the center of the patient's chest in the "high heart" area. This will continue until parents are called to the bedside
  Other Names: Presence
  Arms: Sham Healing Touch Treatment

SUMMARY:
The goal of this study is to assess the benefits of Healing Touch, an energy based therapy on post-operative discomfort and the rate of recovery in children. The aims of this study are to measure the effect of Healing Touch on post-operative: 1) anxiety, 2) emergence agitation/ emergence delirium (EAD), 3) pain, 4) time to wake-up, 5) time to meet PACU's departure criteria, 6.) maladaptive behaviors 2 weeks following surgery & 7)readmissions for complications 2 weeks following surgery.

This is a triple blinded randomized controlled trial with three parallel groups. 240 subjects, ages 3 or 4 will be randomly assigned to receive the usual post-operative care, the usual care plus a post-operative Healing Touch treatment, or the usual post-operative care plus a sham Healing Touch treatment done by an untrained research assistant. The participants & parents, the evaluators, and the principle investigator will be blinded to study group assignment.

DETAILED DESCRIPTION:
ABSTRACT:

Tonsillectomies and adenoidectomies (T&A) are the most commonly performed pediatric surgeries (NIH, 2010). Surgery is understandably anxiety provoking for children and for their families. Research has shown that anxiety influences post-operative recovery (Kain, 2004, 2012; Lynch, 1998; Schisler, 1998; Vaurio, 2006). Anxiety, emergence agitation and emergence delirium (EA/D) and pain during recovery from general anesthesia have been identified as frequent problems in the pediatric population, particularly with younger children (Key, 2010) and these have been related to increases in length of stay. Perioperative stress often has prolonged effects. After surgery, 88% of all children develop new-onset post-operative maladaptive behavioral changes. These changes refer to developmental regression and behaviors that interfere with daily functioning such as general anxiety, nighttime crying, enuresis, separation anxiety, night terrors, temper tantrums etc). Alarmingly, 54% of all children demonstrate maladaptive behaviors 2 weeks following surgery and 20% of these children continue to demonstrate negative behaviors 6 months postoperatively. Research has shown that younger children are at even higher risks (Kain, 2004; Watson, 2003).

Healing Touch is a biofield therapy that has been shown to decrease pain and anxiety in adults (Im, 2009; Jain, 2010) and in premature infants (Hanley, 2008; Im, 2009, Whitley, 2008). For several years Holistic Health Specialist Nurses trained in Healing Touch have been doing Healing Touch in Cincinnati Children's Hospital Medical Center's Post Anesthesia Care Unit (CCHMC's PACU). Nurses anecdotally have noted that patients who receive Healing Touch seem to wake up calmer, often need less pain medication and are less stressful after their surgeries. CCHMC nurses have reported that Healing Touch is especially useful with anxious children and younger children. Healing Touch (HT) is a complementary therapy that is a non-invasive, low-cost therapy without known side effects that can easily be incorporated into post-operative care routines.

The desired study outcomes in the Healing Touch treatment group are:

1. Lower anxiety levels, measured by differences in the Perioperative Adult Child Behavioral Interaction Scale(PACBIS) scores pre & postoperatively. This is a behavioral assessment of the child's coping and distress and the parents positive and negative behavior. Parent will also self evaluated their distress and anxiety. The Healing Touch group will have a lower sympathetic response as measured by preoperative and sequential post-operative B/P, Pulse, Respirations, & pulse oximetry
2. Less emergence agitation and delirium measured by the Pediatric Anesthesia Emergence Delirium (PAED)scores, an observational scale which will be done sequentially once they enter the recovery room
3. Less pain as measured by the Faces, Legs, Activity, Cry, and Consolability (FLACC) scale and significantly less pain medication usage
4. Waking up more slowly once they enter the PACU
5. Shorter length of stay in the PACU, measured by meeting PACU's discharge criteria.
6. Significantly less regression and maladaptive behaviors measured by the Post-Hospital Behavior Questionnaire (PHBQ) 2 weeks following surgery.
7. Fewer readmissions for complications 2 weeks following surgery as identified by family guardian in the 2 week follow up call.

The significance of this study is that its outcomes will add to the body of knowledge about the practice of Healing Touch with children, and may provide evidence substantiating the benefits of Healing Touch on post-operative pediatric patients. This may lead to the incorporation of Healing Touch into pediatric nursing practice. Preschool children are at higher risk for extended stressful responses to surgery, i.e. regression and maladaptive behaviors (Vernon, 1966). Preschoolers have vivid imaginations and magical thinking. They may have trouble telling fantasy from reality. The often develop fears related to new places and experiences and separation from parents. There have been no identified effective supportive measures to improve this protracted stress outcome. Healing Touch may be a tool that can comfort and support this vulnerable population and may be helpful with other hospitalized children.

ELIGIBILITY:
Inclusion Criteria:

Typically developing

* 3 or 4 years old
* elective tonsillectomy with or without adenoidectomy
* o American Society of Anesthesiologist Classification (ASA) I without systemic disease

  o American Society of Anesthesiologist Classification (ASA) II: moderate systemic disease
* Parents speak and write English

Exclusion Criteria:

* Emergency surgery
* have a complicating diagnosis or chronic medical illness
* A history of chronic pain or use of analgesic drugs.
* Familiar or personal history of malignant hyperthermia
* Previous surgeries or hospitalizations
* Parents unable to understand English

Ages: 3 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2013-09; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
1. Anxiety | Day of Surgery (pre and post surgery) & 2 Weeks following Surgery
  1. Perioperative Adult Child Behavioral Interaction Scale (PABCIS) behavioral and self-assessments pre operatively and post-operatively by blinded research assistants. This scale is a behavioral assessment of the child/ adult behavioral interactions in the perioperative period. Parents will be asked to provide self-assessments of their distress in the preoperative and post-operative period. Parents will use Likert scales
  2. Biologic measures: vital signs (B/P, pulse, and pulse oximetry) pre-operatively and sequentially post operatively done by PACU nurses.
  3. 2 Weeks after surgery will do PHBQ (Post Hospital Behavioral Questionaire)to assess childs adaptation

SECONDARY OUTCOMES:
2. Emergence agitation/ emergence delirium | Day of Surgery
  PAED scale done every 5 minutes for the first 30 minutes post op Evaluated from videotape by blinded evaluator

OTHER OUTCOMES:
3. Pain: | Day of Surgery
  1. FLACC pain scores evaluated by bedside nurses when first enter PACU & every 15 min for first hour, every 30 minutes 2nd hour, then every hour until discharge
  2. Assessor, blinded observer will evaluate pain on videotape using modified FLACC scale when subject first arrives in PACU at 15min and 30 minutes and at time when subject meets departure criteria
  3. These FLACC scores done by staff nurses and by assessor will be compared.
  4. Frequency and dose of pain medications (Pre-op/ during surgery/ & post-op)
  5. Type and duration of anesthetic agents will be analyzed.
4. Time to wake up | Day of surgery
  1. From time patient enters the PACU until awake and alert.
  2. Videotape evaluation by blinded observer
5. Length of stay in the PACU: | Day of Surgery
  a. Difference in recorded times-- when subject enters PACU and time subject meets PACU departure criteria as evaluated by PACU nurse. Departure criteria include: Patient is 1. Alert & oriented to place and person and appropriate for age and mental status. 2. Vital signs are stable compared to pre-operative 3. No excessive vomiting as compared to pre-operative 4. Pain is satisfactorily controlled
6. Maladaptive behaviors & ? Has patient needed to be readmitted to hospital for complications | 2 Weeks Post operativly
  1. PHBQ done 2 weeks post operatively (When postoperative pain should no longer be a factor).
  2. This will be done by a phone call to subject's house

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Grace K Rolf, MSN CHTP AHN, Principal Investigator — Cincinnati Childrens
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States